CLINICAL TRIAL: NCT06800391
Title: Metronomic Neoadjuvant Capecitabine and Cyclophosphamide in Huge (PCI>28) Pseudomyxoma Peritonei Patients Candidates to Cytoreductive Surgery (CRS) and Hypertermic Intraperitoneal Chemotherapy (HIPEC)
Brief Title: Metronomic Neoadjuvant Capecitabine and Cyclophosphamide in HUGE Pseudomyxoma Peritonei Patients
Acronym: REVERSE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 135-24; 2024-514329-42-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-25; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Pseudomyxoma Peritonei
Keywords: Pseudomyxoma peritonei; metronomic regimen; capecitabine; cyclophosphamide; cytoreductive surgery; HIPEC; peritoneal cancer index
MeSH Terms: conditions — Pseudomyxoma Peritonei | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Capecitabine will be taken orally at dose of 1250 mg/m2 /day (625 mg/m2 BID), continuous daily dosing. Cycles are to be repeated every 28 days for a total of 6 cycles.
  Cyclophosphamide 50 mg/day continuous daily dosing. Cycles are to be repeated every 28 days for a total of 6 cycles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capecitabine and Cyclophosphamide (Experimental): Capecitabine (1250 mg/m2 /day) and Cyclophosphamide (50 mg/day) continuous daily dosing.
  Cycles are to be repeated every 28 days for a total of 6 cycles.
  Interventions: Combination Product: Capecitabine 1250 mg/m2 /day - Cyclophosphamide 50Mg/day

INTERVENTIONS:
Combination Product: Capecitabine 1250 mg/m2 /day - Cyclophosphamide 50Mg/day — Capecitabine (1250 mg/m2 /day) and Cyclophosphamide (50 mg/day) continuous daily dosing. Cycles are to be repeated every 28 days for a total of 6 cycles.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of neoadjuvant capecitabine and cyclophosphamide treatment in patients affected by huge Pseudomyxoma peritonei (PMP) (peritoneal cancer index >28). Treatment consists of metronomic (low-dose medication for a prolonged time) of capecitabine plus cyclophosphamide for 6 months followed by standard of care cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC). The main question the trial aims to answer is which is the proportion of patients with complete cytoreduction at CRS/HIPEC after neoadjuvant metronomic approach with oral capecitabine and cyclophosphamide in patients affected by huge PMP.

DETAILED DESCRIPTION:
Mucinous neoplasms are the most common appendiceal tumors, and the most common cause of Pseudomyxoma peritonei (PMP). The term PMP defines a clinical syndrome characterized by progressive accumulation of mucinous material within the abdominal-pelvic cavity, ultimately leading to patient death due to local-regional progression of the disease. The upfront cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) is regarded as standard treatment for PMP.

However, not every PMP patient benefit from upfront CRS and HIPEC. A proportion of patients could be inoperable due to a lack of clinical conditions for clinical deterioration or comorbidites contra-indicating surgery, or an unresectable disease at the diagnosis. Up to 32% of cases could be present the so-called huge PMP (peritoneal cancer index >28), where the proportion of patients with complete cytoreduction is low of their entire cohort of PMP patients. Moreover, CRS in huge PMPs generally requires very extensive surgical maneuvers such as total gastric or total colon resection. Hence, the patients suffer from a significant impact on postoperative quality of life due to nutritional issues.

Preoperative systemic chemotherapy might be an option for such advanced cases, as it can possibly reduce the tumor burden, allowing less extensive surgery with less visceral resections. Systemic treatment regimens are associated with relevant toxicity and highcosts. Metronomic schedules might be preferred because of their favorable safety profileand antiangiogenic and immunomodulatory properties.

In unresectable or progressive PMP, a single-center prospective uncontrolled trial showed the safety and promising activity results of a continuous metronomic regimen with capecitabine with cyclophosphamide. At a median follow-up of 22.4 months, median progression-free survival was 9.5 months, and the 1-year overall survival rate was 73.7%. Overall, the disease control rate was 87%, and 6 (27%) patients achieved disease control ≥12 months.

On this basis, a phase II, mono-institutional, single arm trial was designed, evaluating neoadjuvant metronomic capecitabine and cyclophosphamide in patients affected by huge Pseudomyxoma peritonei who are potentially candidates to cytoreductive surgery and HIPEC. The goal of the present study is to evaluate the surgical and oncological outcomes of neoadjuvant metronomic approach with oral capecitabine and cyclophosphamide in patients affected by huge PMP.

In details, after the identification of patients affected by PMP, the measurement of peritoneal cancer index will be assessed by chest and abdominal CT scan at the staging phase. Only patients with PCI>28 will be recruited regardless of resectability. Once enrolled, the patients will receive staging laparoscopy in order to confirm the histological diagnosis, to accurately stage the disease with the surgical PCI, to be compared with the radiological PCI for accuracy evaluation, and to collect material for the translational analyses. Then the patients will receive a continuous treatment schedule of oral metronomic chemotherapy with capecitabine 1250 mg/m2/day (625 mg/m2 BID) continuously with cyclophosphamide 50 mg/day continuously, for a total of 6 four-weekly cycles. At the completion of the cycles, the patients will be restaged and, as long as they are considered operable, they will be submitted to standard of care cytoreductive surgery/HIPEC, in order to define the reaching of the primary endpoint of completeness of cytoreduction. A total number of 31 patients are planned to be included in the study according to the statistical design.

ELIGIBILITY:
Inclusion Criteria:

* Clinical/Histological diagnosis of pseudomyxoma peritonei (PMP);
* Peritoneal Cancer Index (PCI >28) assessed by chest and abdominal CT scan at the staging phase;
* Age >= 18 years and <76 years;
* Performance Status (ECOG <2);
* Adequate organ function including the following:
* Adequate bone marrow reserve: WBC count >3.0x109/L, absolute neutrophyl count >1.5x109/L, platelet count >100x109/L, and hemoglobin >10 g/dL;
* Hepatic: bilirubin < 1.5 times the ULN, alkaline phosphatase, aspartate transaminase, and alanine transaminase < 2.5 x UL;
* Renal: Creatinine clearance >50 mL/min or serum creatinine <1.5 x UNL;
* Patients compliance and geographic proximity that allows for adequate follow-up;
* Patients must sign an informed consent document (ICD);
* Male and female patients with reproductive potential must use an approved contraceptive method;

Exclusion Criteria:

* Peritoneal Cancer Index (PCI ≤28) assessed by chest and abdominal CT scan at the staging phase;
* DPD deficiency;
* Previous systemic chemotherapy and/or biological therapy;
* Administration of other experimental drugs during the study Pregnancy and breast-feeding;
* Serious or uncontrolled medical pathologies or active infections that would jeopardize the possibility of receiving the investigated treatment;
* Disorders that could influence the absorption of capecitabine (e.g. malabsorption), intestinal occlusion, Crohn's disease or ulcerative colitis;
* Psychiatric disorders, neurologic disease or other conditions that would make it impossible to comply with the protocol procedures;
* Positive anamnesis with regard to other neoplastic diseases except for the ones that have been cured for more than 5 years.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with complete cytoreduction after neoadjuvant metronomic approach with oral capecitabine and cyclophosphamide in patients affected by huge PMP. | 6-8 months from the start of treatment
  Use of Completeness of Cytoreduction score to evaluate the radicality of Cytoreductive Surgery. Patients with a residual disease <2.5 mm will be considered completely cytoreduced, otherwise incompletely cytoreduced.
  "Completeness of Cytoreduction Score" ranging from the best cc-0: no peritoneal nodule was seen, afterwards cc-1,tumor nodules persisting after cytoreduction are less than 2.5 mm in diameter, then cc-2, tumor nodules persisting after cytoreduction are between 2.5 mm and 2.5 cm in diameter to the worst cc-3, tumor nodules persisting after cytoreduction are greater than 2.5 cm

SECONDARY OUTCOMES:
Radiological objective tumor response rate. | Performed at baseline and 16 weeks from the start of treatment.
  Objective tumor response rate will be defined by two independent radiologists by means of CT (computed tomography) scans. Tumour response will be determined semiquantitatively as either stable, reduced or progressed.
Conversion rate | 6-8 months from the start of treatment
  Conversion rate will be calculated dividing the number of resectable cases after the neoadjuvant chemotherapy by the number of resectable cases before neoadjuvant chemotherapy. Resectability will be evaluated with CT scans using Bouquot et al. methodology.
Downsizing of the tumor measured by surgical Peritoneal Cancer index (PCI). | Performed after 16 weeks.
  Downsizing of the tumor will be measured at the time of staging laparoscopy and CRS using Peritoneal Cancer Index (PCI). Peritoneal cancer index (PCI) ranging from the best 0 to the worst 39.
Safety and tolerability of neoadjuvant metronomic chemotherapy. | 6-8 months.
  Incidence of Treatment-Emergent Adverse Event will be measured using NCI-CTCAE v5.
Major complications (NCI-CTCAE v5) associated with CRS and HIPEC | 30 days after surgery.
  Major complications associated with CRS and HIPEC will be measured using NCI-CTCAE v5.
Quality of life EQ-5D-5L | Before/after neoadjuvant metronomic chemotherapy, and 30 days after the surgery.
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument. EuroQol EQ-5D-5L. The EQ-5D-5L uses for first 5 questions qualitative multiple choice answers with NO SCALE. For the last questions, a score from 0 to 100 indicates from the worst to the best outcome.
Progression-free survival | After 24 months.
  Progression-free Survival (PFS) is the time between the date of chemotherapy commencement and the date of Disease-Progression or Death, whichever occurs first.
Overall Survival. | After 48 months.
  Overall Survival (OS) is the time between the date of chemotherapy commencement and date of Death or last follow up.
Quality of life EORTC-QLQ-C30 | Within 30 days after the date of surgery.
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument. EORTC QLQ-C30 For questions 1-28 of EORTC QLQ-C30 a 4-point scale is used. It scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit")and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome. For the questions 29 and 30 of EORTC QLQ-C30 a 7-points scale is used. It scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.

OTHER OUTCOMES:
Effect of neoadjuvant metronomic chemotherapy on the immunocompetence of tumor microenvironment | Through the study completion, an average of 3 years
  Conduction of biological studies with exploratory nature and therefore without the possibility to be categorized according to specific scale of range.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Raimondi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy